CLINICAL TRIAL: NCT03221088
Title: Pegylated Somatropin (PEG Somatropin) in the Treatment of Children With Idiopathic Short Stature: A Controlled, Prospective, Randomized, Multicenter Phase-II Study With An Untreated Control Group.
Brief Title: A Study of PEG-somatropin in the Treatment of Children With Idiopathic Short Stature
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other); The First Hospital of Jilin University (Other); Affiliated Hospital of Jiangnan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Children's Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 033 CT-one year
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Dwarfism
MeSH Terms: conditions — Dwarfism | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jintrolong® low dose group (Experimental): PEG-rhGH Injection (27IU/4.5mg/0.5ml/bottle) 0.1 mg/kg/w by subcutaneous injection for 52 weeks.
  Interventions: Drug: Jintrolong® low dose group; Drug: Jintrolong® high dose group
- Jintrolong® high dose group (Experimental): PEG-rhGH Injection (27IU/4.5mg/0.5ml/bottle) 0.2 mg/kg/w by subcutaneous injection for 52 weeks.
  Interventions: Drug: Jintrolong® low dose group; Drug: Jintrolong® high dose group
- Negative control group (No Intervention): Untreated Control Group

INTERVENTIONS:
Drug: Jintrolong® low dose group — PEG-somatropin 0.1mg/kg/wk by weekly subcutaneous injection for 52 weeks.
  Other Names: PEG-somatropin
  Arms: Jintrolong® high dose group; Jintrolong® low dose group
Drug: Jintrolong® high dose group — PEG-somatropin 0.2 mg/kg/wk by weekly subcutaneous injection for 52 weeks.
  Other Names: PEG-somatropin
  Arms: Jintrolong® high dose group; Jintrolong® low dose group

SUMMARY:
This study aims to explore the optimal dose of pegylated recombinant human growth hormone (PEG-rhGH) injection to treat children with idiopathic short stature (ISS), evaluate its safety and efficacy, and provide scientific and reliable evidence for the medication dosage in Phase III clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Boys are between 4 and 9 years of age and girls are between 4 and 8 years of age.
* Height <-2 SD for chronological age.
* Growth velocity<5.0 cm/yr.
* GH peak concentration ≥10.0 ng/mL in two different stimulation tests.
* The difference of bone age (BA) and chronological age (CA) is within -2 to +2.
* IGF-1 concentration is between -2 SDS to +2 SDS.
* Prepubertal Status(Tanner Stage I).
* Birth weight within the normal range.
* Growth hormone treatment-naive.
* Subjects are willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, to sign informed consent.

Exclusion Criteria:

* Subjects with abnormal liver and kidney functions (ALT > upper limit of normal value; Cr > upper limit of normal value).
* Subjects are positive for anti-HBc, HbsAg or HbeAg in Hepatitis B virus tests.
* Subjects with known highly allergic constitution or allergy to investigational product or its excipient.
* Subjects with systemic chronic disease and immune deficiency.
* Patients diagnosed with tumor.
* Patients with mental disease.
* Patients with other types of abnormal growth and development.

  1. Growth hormone deficiency (GHD) (confirmed by GH stimulation test);
  2. Turner syndrome (confirmed by karyotype test of girls);
  3. Noonan syndrome (hypertelorism, pectus carinatum, hypophrenia, frequently with skin disease and congenital heart disease, missense mutation of the protein tyrosine phosphatase, non-receptor type 11 (PTPN11) gene on chromosome 12 for half of the patients, for both male and female patients);
  4. Laron sydrome (confirmed by IGF-1 generation test);
  5. Small for gestational age ( the birth height or weight is below the tenth percentile or 2 SD, with catch-up growth uncompleted at 2 years old).
* Growth disorders caused by malnutrition or hypothyroidism (thyroid function test).
* Congenital skeletal abnormalities or scoliosis, claudication.
* Subjects with impaired glucose regulation (IGR) (including impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) ) or diabetes).
* Subjects with abnormal electrolyte, blood gas analysis (vein), creatine kinase.
* Subjects who took part in other clinical trials within 3 months.
* Subjects who received medications which may interfere GH secretion or GH function, or other hormones within 3 months (such as sex steroids, glucocorticoids, etc.).
* For patients with potential high tumor risks such as tumor markers exceed normal range and some other relative information, they may be excluded from the treatment.
* Other conditions which is inappropriate for this study in the opinion of the investigator.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Height Standard Deviation Score for Chronological Age (ΔHtSDSCA) | Baseline，52 weeks
  Change in Height Standard Deviation Score for Chronological Age (ΔHtSDSCA) from Baseline to 52 weeks；ΔHtSDSCA=(height Yx - reference mean for CA Yx) / reference SD for CA Yx (Yx refers to the height value at particular timepoint x)

SECONDARY OUTCOMES:
Change in Annualized Height Velocity | Baseline，52 weeks
  Annualized Height Velocity=12×(Height Yx - Height at Baseline)/(Date of Yx - Date of Baseline) (Yx refers to the height value at particular timepoint x)
Change in Bone Maturation | Baseline，52 weeks
  Bone Maturation=(BA Yx-BA at Baseline)/(Date of Yx - Date of Baseline) (Yx refers to the BA value at particular timepoint x)
Change in IGF-1 Standard Deviation Score (IGF-1 SDS) | Baseline，52 weeks
  GF-1 SDS=(IGF-1 Yx - reference mean for CA Yx) / reference SD for CA Yx (Yx refers to the IGF-1 value at particular timepoint x)
IGF-1/IGFBP-3 molar ratio at 52 weeks | Baseline，52 weeks
  IGF-1/IGFBP-3 molar ration=[IGF-1(ng/ml)/7.6]/[IGFBP-3 (ng/ml)/25.75]

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Principal Investigator — Department of Pediatrics of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (7):
- China (7):
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shanghai Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's Hospital, Shanghai